CLINICAL TRIAL: NCT04511520
Title: Clinical Efficacy of Personalized Exercise Program and an Inhibitor of Fatty Acid β-oxidation in Rehabilitation of Patients With Atrial Fibrillation After Primary Radiofrequency Ablation of Pulmonary Venous Orifices
Brief Title: Efficacy of Personalized Exercise Program and Trimetazidine in Rehabilitation of Patients After RFA of AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PTAF02-02/13
Record Dates: First submitted 2020-06-10; First posted 2020-08-13 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: rehabilitation; atrial fibrillation; physical training; radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Trimetazidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physical training (Experimental): Integrated Rehabilitation consisting of exercise training (minimum 3 times a week for a total of 6 months)
  Interventions: Other: Physical training program
- Trimetazidine (Experimental): Treatment of trimetazidine in addition to standart therapy
  Interventions: Drug: Trimetazidine
- Control (No Intervention): Standard follow-up at the participating heart center

INTERVENTIONS:
Other: Physical training program
  Arms: Physical training
Drug: Trimetazidine
  Other Names: fatty acids beta-oxidation inhibitor
  Arms: Trimetazidine

SUMMARY:
Atrial fibrillation (AF) is one of the most common forms of heart rhythm disorder in patients with cardiovascular diseases. The choice of treatment for AF is a complex problem, depending on the form (paroxysmal, persistent, permanent) of AF, clinical manifestations of cardiac arrhythmias, associated diseases, the effectiveness of antiarrhythmic drugs. The accumulated data to date indicate an efficacy of the method of radiofrequency ablation (RFA) in the treatment of the paroxysmal form of AF. The RFA procedure does not eliminate the pathological processes that take place during developed AF. This dictates the need to develop and test new technologies and physical rehabilitation programmes for patients. The positive clinical effects of physical rehabilitation programmes based on moderate-intensity exercises are well known. The search for drugs capable of improving the results of RFA for AF in patients becomes urgent. This creates the prerequisites for the study of the clinical efficacy of trimetazidine MV in the rehabilitation of patients with cardiac diseases who underwent treatment of AF with RFA, which will optimize the management of such patients in the inpatient and outpatient setting.

DETAILED DESCRIPTION:
The study is interventional (Clinical Trial), randomized in parallel groups. Enrollment: 72 participants.

The 72 male patients were randomized in 3 groups. In 1st group (control) patients were taken antiarrhythmical drugs and anticoagulants. They did only usual activity without walking. Patients in 2nd group were taken antiarrhythmical drugs and anticoagulants, participated in rehabilitation programme. Twice a week they came in clinical center to engage in physical training with an instructor. The programe was lasted for 6 months. Also patients did they usual physical activity, practiced walking. Patients in 3rd group were taken antiarrhythmical drugs and anticoagulants, selective inhibitor of fat acids oxidation for 6 months. They did only usual activity without walking.

The examination was carried for all 72 patients. Before RFA patients took blood tests, performed echocardiography, completed psychological questionnaires. After 3 days they took blood tests, performed 6-minute walk testing, ECG monitoring, completed psychological questionnaires. One month after RFA patient performed veloergometry testing. Three months after RFA the performed 6-minute walk testing, ECG monitoring, took blood tests, completed psychological questionnaires. Six months after RFA patients took blood tests, performed echocardiography, 6-minute walk testing, ECG monitoring, veloergometry testing, completed psychological questionnaires. Onward was a follow up period for 6 months. At the time point of 12 months patients took blood tests, performed echocardiography, ECG monitoring, veloergometry testing, completed psychological questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* treated for atrial fibrillation with radiofrequency ablation
* cardiac disease
* providing written informed consent

Exclusion Criteria:

* Congenital and acquired heart defects.
* Acute coronary syndrome (unstable angina, myocardial infarction), myocardial revascularization during the previous 6 months
* Transient ischemic attack, stroke in history.
* Arterial hypertension (BP ≥160/100 мм. рт. ст.)
* The risk of thromboembolic complications on a scale CHA2DS2-VASc> 2
* Risk of hemorrhagic complications of anticoagulant therapy (HAS-BLED> 3 points on the scale).
* Complications after RFA.
* Chronic heart failure above III FC (NYHA), ejection fraction (EF) <40%.
* Acute thrombophlebitis, complicated forms of varicose veins (thrombophlebitis, phlebothrombosis).
* Pronounced atherosclerosis of peripheral arteries (intermittent claudication), requiring surgical intervention.
* Violation of conductivity: AV-blockade 2-3 degrees, complete blockade of the bundle of the His bundle
* The presence of an implanted pacemaker pacemaker / pacemaker with a resynchronization function/cardioverter-defibrillator)
* Conduct RFA on AF earlier.
* The presence of a history of syncopal states.
* Diabetes mellitus type 1 and 2 in the stage of decompensation.
* Acute conditions: infection, exacerbation of chronic diseases in a period of less than 1 month prior to the study; severe injury, surgical interventions other than RFA for a period of less than 2 months from the start of the study
* Renal failure (creatinine levels above 300 µmol / L or 3.5 mg / dL).
* Patient's refusal to participate in the study
* Alcohol and drug abuse.
* Peptic ulcer and duodenal ulcer in history.
* Obesity, body mass index (BMI) ≥40 kg / m2
* Intake of Trimetazidine MB and its analogues for 3 months. before inclusion in research.
* The presence of any disease that, according to the doctor, prevents the inclusion of the patient in the study.
* unable to understand study instructions
* with considerable illness in the musculoskeletal system or with physical disability, which complicates exercise training

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol
Time Frame: until December 2020
Access Criteria: study protocol will be available upon request

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no significant study events
Groups:
- Physical Training: Integrated Rehabilitation consisting of exercise training (minimum 3 times a week for a total of 6 months)
  Physical training program
- Trimetazidine: Treatment of trimetazidine in addition to standard therapy
  Trimetazidine
Period: Overall Study
Arm/Group | Physical Training | Trimetazidine | Control
Started | 24 | 24 | 24
Completed | 24 | 24 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Trimetazidine: Treatment of trimetazidine in addition to standart therapy
  Trimetazidine
- Total: Total of all reporting groups
Arm/Group | Physical Training | Trimetazidine | Control | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (8.5) | 56.4 (8.1) | 55.0 (9.8) | 56.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 24 | 24 | 24 | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation Recurrence
Description: Number of participants with reccurrence of atrial fibrillation after RFA
Time Frame: From RFA to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Training | Trimetazidine | Control
Number analyzed (Participants) | 24 | 24 | 24
Participants | 2 | 3 | 7

2. Primary Outcome: Atrial Fibrillation Recurrence
Description: Number of participants with recurrence of atrial fibrillation after RFA
Time Frame: From 3 months to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Physical Training: Integrated Rehabilitation consisting of exercise training (minimum 3 times a week for a total of 6 months)
  Physical training programme
Arm/Group | Physical Training | Trimetazidine | Control
Number analyzed (Participants) | 24 | 24 | 24
Participants | 1 | 2 | 4

3. Primary Outcome: Atrial Fibrillation Recurrence
Description: Number of participants with recurrence of atrial fibrillation after RFA
Time Frame: From 6 months to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Training | Trimetazidine | Control
Number analyzed (Participants) | 24 | 24 | 24
Participants | 6 | 6 | 9

ADVERSE EVENTS:
Arm/Group | Physical Training | Trimetazidine | Control
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes